CLINICAL TRIAL: NCT02701335
Title: Neural Manual vs. Robotic Assisted Mobilization to Improve Hand Range of Motion and Reduce Pain Hypersensitivity in Hand Osteoarthritis: a Randomized Controlled Trial
Brief Title: Manual Therapy for Hand Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Project Code:GR-2013-02358472
Record Dates: First submitted 2016-02-27; First posted 2016-03-08 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hand Osteoarthritis
Keywords: Osteoarthritis; Hand; Rehabilitation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Neural mobilization and standardized exercise . 12 sessions over 4 weeks (3 sessions per week).
  Interventions: Device: Neural mobilization; Device: Standardized exercise
- Control group (Active Comparator): Gloreha device and standardized exercise. 12 sessions over 4 weeks (3 sessions per week).
  Interventions: Device: Gloreha device; Device: Standardized exercise

INTERVENTIONS:
Device: Neural mobilization — The first 6 exercises consist of active range of motion movements of the hand designed to improve joint flexibility. The remaining 3 exercises are designed to strengthen grip and pinch by using a non-latex polymer ball: the Thera-Band Hand Exerciser (The Hygenic Corporation, Akron, OH) Subjects began with 10 repetitions the first 4 sessions, progressed to 12 repetitions the next 2 sessions, then 15 (2 sessions), and finally 20, if able, during the last sessions.
  Arms: Experimental group
Device: Gloreha device — Robotic assisted passive mobilization.
  Arms: Control group
Device: Standardized exercise — 9 exercises: active range of motion, strengthen grip and pinch

SUMMARY:
Osteoarthritis (OA) of the hand is a major cause of pain and functional limitation, central sensitization of pain can be one of the causes: this hypothesis opens avenues for research in the modulation of pain pathways. The peripherally directed therapies may modulate pain perception bilaterally. This hypothesis opens avenues for future research in the modulation of pain pathways, perhaps offering targets to optimize peripheral manual and physical therapies for pain management in hand OA.

Several studies have reported the outcomes of multimodal approach to central sensitization evaluated by generalized pressure pain hypersensitivity in patients with carpometacarpal (CMC) OA. Neurodynamic techniques are a form of manual therapy directed to the neural structures through positioning and movement of multiple joints. Recent technologies have facilitated the use of robots as tools to assist patients in the rehabilitation process thus maximizing patient outcomes. These robotic tools assist the patient with carrying out exercise protocols, optimal for the activity of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the dominant hand. To be included in the study, the subjects need to have a history of repetitive use of their dominant hand (eg, ex-factory worker) and a diagnosis of hand OA in the dominant hand, according on radiographic findings.

Exclusion Criteria:

* If they score greater than 6 points on the Beck Depression Inventory (BDI) or more than 30 points in the State Trait Anxiety Inventory (STAI). Patients with a medical history of carpal tunnel syndrome, surgical interventions to the hand, DeQuervain's tenosynovitis, or with degenerative or non-degenerative neurological conditions in which pain perception is altered will be excluded. None of the individuals in this study will have received prior interventions for hand OA.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from Pain intensity at 3 months | baseline, immediately post-intervention, and at 1- and 3-month post-interventions, Baseline up to 5 minutes.
  visual analogue scale
Change from QuickDASH questionnaire at 3 months | baseline, immediately post-intervention, and at 1- and 3-month post-interventions Baseline, up to 5 minutes.
  will be used to measure upper extremity function
Change from Pressure Pain Thresholds (PPT) at 3 months | Baseline and immediately post-interventionand, at 1- and 3-month post-interventions.
  is a quantitative sensory test of tissue sensitivity and it is defined as the minimal amount of pressure that produces pain, measured via a pressure algometer. PPT will be assessed bilaterally over the hand (first CMC at the center of the anatomical snuffbox, and unciform apophysis of the hamate bone), the C5-C6 zygapophyseal joint, the median, ulnar and radial nerves, and tibialis anterior muscle by an assessor blinded to the subjects condition.

SECONDARY OUTCOMES:
Motor conduction velocity | Baseline up to 5 minutes
Range of Motion | Baseline up to 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Hugo Villafañe, Piossasco, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersini P, Valdes K, Cantero-Tellez R, Cleland JA, Bishop MD, Villafane JH. Effects of Neurodynamic Mobilizations on Pain Hypersensitivity in Patients With Hand Osteoarthritis Compared to Robotic Assisted Mobilization: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2021 Feb;73(2):232-239. doi: 10.1002/acr.24103. Epub 2021 Jan 3. PMID 31675184